CLINICAL TRIAL: NCT04201158
Title: A Comparison of Activities of Daily Living, Physical Fitness and Quality of Life in Obese and Healthy Adolescents
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO19/60
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Obesity, Childhood; Healthy
Keywords: Physical Fitness; Exercise Capacity; Activities of Daily Living; Quality of Life
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese Group (Girl): Diagnosed with the obesity according to body mass index reference system, being 10-18 years old, being volunteer for the research and able to walk and cooperate are the inclusion criteria.Diagnosed with a neurological disease or another clinical diagnosis that may affect the cognitive state, musculoskeletal and neurological disease, symptomatic heart disease, lung disease, diabetes, hypertension and malignant disease, which may affect the performance of exercise and using the drug that affects appetite and weight are the exclusion criteria.
  Interventions: Diagnostic Test: Exercise Capacity
- Obese Group (Boy): Diagnosed with the obesity according to body mass index reference system, being 10-18 years old, being volunteer for the research and able to walk and cooperate are the inclusion criteria. Diagnosed with a neurological disease or another clinical diagnosis that may affect the cognitive state, musculoskeletal and neurological disease, symptomatic heart disease, lung disease, diabetes, hypertension and malignant disease, which may affect the performance of exercise and using the drug that affects appetite and weight are the exclusion criteria.
  Interventions: Diagnostic Test: Exercise Capacity
- Control Group (Girl): Being normal weight according to body mass index reference system, being 10-18 years old, being volunteer for the research and able to walk and cooperate are the inclusion criteria. Having comorbidities which may affect exercise performance and other physical tests, diagnosed with the cardiovascular problems, musculoskeletal and neurological diseases, cognitive or motor limitation or other chronic diseases are exclusion criteria.
  Interventions: Diagnostic Test: Exercise Capacity
- Control Group (Boy): Being normal weight according to body mass index reference system, being 10-18 years old, being volunteer for the research and able to walk and cooperate are the inclusion criteria. Having comorbidities which may affect exercise performance and other physical tests, diagnosed with the cardiovascular problems, musculoskeletal and neurological diseases, cognitive or motor limitation or other chronic diseases are exclusion criteria.
  Interventions: Diagnostic Test: Exercise Capacity

INTERVENTIONS:
Diagnostic Test: Exercise Capacity — Modified Shuttle Walk Test

SUMMARY:
It is known that activities of daily living, physical fitness, exercise capacity and quality of life are affected by the obesity. It is aimed to determine the effects obesity on daily living activities, physical fitness, exercise capacity and quality of life in obese adolescents compared to healthy subjects in this study. The relationship between these parameters and the activities of daily living which are less studied in obese adolescents will be evaluated.

DETAILED DESCRIPTION:
Obesity among children, adolescents and adults has emerged as one of the most serious public health problems in the 21st century. There has been a significant decrease in the exercise capacity, physical fitness and activities of daily living of children and adolescents with the increase in the prevalence of obesity over the last decade. Obesity can cause not only health problems but also psychological effects. This situation have negative effects on the quality of life. The effect of these parameters on healthy individuals and obese adolescents will be demonstrated by this study and will guide the rehabilitation of obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

Healthy group:

* Being normal weight according to BMI reference system,
* Being between the ages of 10-18 and volunteer to participate in the research,
* Being able to walk and cooperate

Obese Group:

* Obesity diagnosis according to BMI reference system,
* Being between the ages of 10-18 and volunteer to participate in the research,
* Being able to walk and cooperate.

Exclusion Criteria:

Healthy Group:

* Comorbidities that may affect exercise performance and other physical tests,
* Having cardiovascular problems, musculoskeletal and neurological disease,
* Having cognitive or motor limitation or other chronic diseases.

Obese Group:

* Having a neurological disease or other clinical diagnosis that may affect cognitive status,
* Having musculoskeletal and neurological diseases, symptomatic heart disease, lung disease, diabetes, hypertension and malignant disease that may affect exercise performance,
* Using medication that affects appetite and weight.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — 15 obese adolescents, 15 obese adolescent adolescents and 15 healthy female adolescents and 15 healthy male adolescents compatible with age and sex will be recruited from obese adolescents according to the BMI reference system.
Study Population: 15 obese adolescents, 15 obese adolescent adolescents and 15 healthy female adolescents and 15 healthy male adolescents compatible with age and sex will be recruited from obese adolescents according to the BMI reference system.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
The Modified shuttle walk test. | February 2019-February 2020
  Maximal exercise capacity

SECONDARY OUTCOMES:
Waist circumference, Abdominal circumference, Ratio of waist to hip | February 2019-February 2020
  Antropometric measurements
Hand grip strength by hand dynamometer (Jamar). | February 2019-February 2020
  Peripheral Muscle Strength
the Glittre Activities of Daily Living (ADL) Test. | February 2019-February 2020
  Activities of daily living
the Munich Physical Fitness Test-MFT | February 2019-February 2020
  Physical Fitness
Modified push-ups, shuttles and squats as possible for 30 seconds | February 2019-February 2020
  Peripheral muscle endurance
The Pediatric Outcomes Data Collection Instrument (PODCI) | February 2019-February 2020
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Iskenderoglu, Physical Therapist, Study Chair — Hacettepe University; Deniz Inal Ince, Professor, Study Chair — Hacettepe University; Melda Saglam, Associate Professor, Study Chair — Hacettepe University; Naciye Vardar Yagli, Associate Professor, Study Chair — Hacettepe University; Hazal Sonbahar Ulu, MSc, Study Chair — Hacettepe University; Melis Pehlivanturk Kizilkan, MD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided